CLINICAL TRIAL: NCT01641484
Title: Study Evaluating Predictive Value of Local Control at 19.8 (MRI and TEP Scan) for Patient With Stade I to IIIB Cervix Carcinoma Treated by Radiotherapy
Brief Title: Study of a Predictor for Cervix Cancer
Acronym: ANOXICOL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: unreached recruitment objectives
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ANOXICOL-1102
Record Dates: First submitted 2012-07-06; First posted 2012-07-16 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Cervix Cancer; Oncology
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- local control 19.8Gy (Experimental): local control at 19.8 Gy, at Day 14
  Interventions: Procedure: local control at 19.8Gy

INTERVENTIONS:
Procedure: local control at 19.8Gy — Day 14, full body TEP and pelvis MRI

SUMMARY:
Non operated cervix cancer are usually treated by radio-chemotherapy. Non control local rate is inexplicably close to 30%. However, important volume of those tumors and their hypoxia degree induce phenomenon of pathologic angiogenesis, explaining these therapeutic failures.

Persistence of tumor hypoxia could be a predictive factor of local control

DETAILED DESCRIPTION:
HPV linked cervix cancer is the second most prevalent form of female cancer. It's also the leading cause of death by cancer in Asia, South America and Africa. Hopefully, screening program lead to a 50 % of mortality reduction during the past 40 years. Classic therapeutic strategy consists of external pelvic radiation therapy associated with chemotherapy and followed by brachytherapy. Curative surgical removal is realized 4 to 6 weeks after radiation therapy. However relapse rate is frequent (20 to 30%). Biological mechanisms involved in this high relapse rate are not understood.

Nevertheless, it is suggest that initial hypoxia of cervix tumor during 20 Gy radiation therapy is a pejorative prognostic factor. At the opposite, the amelioration of tumor vascularisation during 20 Gy radiation therapy is a positive prognostic factor. It's possible that an amelioration of hypoxia lead to lesser tumor resistance to radiotherapy. However such possibility has to be test during clinical trial.

Thus, the objective of ANOXICOL study is to evaluate the predictive value of persistent hypoxia, during 20 Gy radiation therapy associated with chemotherapy, for local control of cervix cancer.

ELIGIBILITY:
Inclusion Criteria:

* cervix epidermoid cancer or adenocarcinoma : I to IIIB
* treatment by radiochemotherapy
* ECOG ≤ 1
* social and psychological compliance for standard treatment of radiochemotherapy for cervix carcinoma
* patient affiliated to health insurance system
* signed informed consent

Exclusion Criteria :

* contraindication to chemoradiotherapy
* resequable cervical cancer
* para-aortic metastases histologically proven
* inability to perform an abdominal MRI or a PET Scan
* contraindications related to MRI: pacemaker, vascular clip, and all devices incompatible with the electromagnetic field generated by MRI
* unbalanced diabete
* administration of EPO
* transfusion within 3 days before the first biopsy
* creatinine clearance under 60 mL / min;
* ANC <1500 / mm3 and Platelets <120,000 / mm3
* neuropathy, diabetes (fasting glucose greater than 140 mg / l) or any other condition that strongly contraindicates concomitant chemotherapy with radiotherapy
* sigmoid diverticulitis, Crohn's disease or systemic disease, collagenose

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
change from baseline of value of persisting hypoxia at day 14 | Baseline, Day 14
  dynamic MRI : tumor volume, intensity of contrast enhancement (Ktrans and SI10 measurement) TEP scan : metabolic intensity, SUV measurement comparison of biopsie negativity

SECONDARY OUTCOMES:
safety | baseline, Day 14, Day 45, Day 120
  NCI CTCAE v 4.0
MRI and TEP local control evaluation | 4 months
impact of tumor hypoxia on necrosis appearance | Day 45 and Day 120
  necrosis quantification from biopsies
correlation between biomarkers of tumor hypoxia evolution and local control | baseline, Day 14, Day 45 and Day 120
  evaluate necrosis appearance as a proxy to local control

CONTACTS AND LOCATIONS:
Overall Officials: Nickers Philippe, MD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Oscar Lambret Center, Lille, France

IPD SHARING:
Plan to Share IPD: No